CLINICAL TRIAL: NCT04725721
Title: Testing FIRST in Youth Outpatient Psychotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, John Weisz, Professor, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB20-1875
Record Dates: First submitted 2021-01-10; First posted 2021-01-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Depression; Trauma; Behavior Problem
Keywords: anxiety; depression; trauma; behavior problems; youth; mental health; emotion regulation
MeSH Terms: conditions — Anxiety Disorders; Depression; Wounds and Injuries; Mental Disorders; Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIRST (Experimental): FIRST is built upon five empirically supported principles of change (ESPCs-i.e., feeling calm, increasing motivation, repairing thoughts, solving problems, trying the opposite). Each principle can be applied to treatment of problems spanning depression, anxiety (including OCD and PTS), and conduct problems-thus encompassing a majority of the youths seen in outpatient care. Its design addresses breadth of problem coverage, youth comorbidity, and flux in youth treatment needs during episodes of care. It is used in conjunction with performance feedback via a web-based tracking system that gives clinicians weekly data on youth treatment response. FIRST has treatment and training efficiency, and efficient clinician skill-building is supported by group consultation.
  Interventions: Behavioral: FIRST
- Usual Care (Active Comparator): Treatment in the usual care (UC) condition will use the clinical procedures therapists consider appropriate and believe to be effective.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: FIRST — FIRST is built upon five empirically supported principles of change (ESPCs-i.e., feeling calm, increasing motivation, repairing thoughts, solving problems, trying the opposite). Each principle can be applied to treatment of problems spanning depression, anxiety (including OCD and PTS), and conduct problems-thus encompassing a majority of the youths seen in outpatient care. Its design addresses breadth of problem coverage, youth comorbidity, and flux in youth treatment needs during episodes of care. It is used in conjunction with performance feedback via a web-based tracking system that gives clinicians weekly data on youth treatment response. FIRST has treatment and training efficiency, and efficient clinician skill-building is supported by group consultation.
  Arms: FIRST
Behavioral: Usual Care — Treatment in the usual care (UC) condition will use the clinical procedures therapists consider appropriate and believe to be effective.
  Arms: Usual Care

SUMMARY:
The study will compare the impact FIRST (a transdiagnostic treatment built upon five empirically supported principles of change) versus usual care outpatient psychotherapy on youths' mental health outcomes and a candidate mechanism of change: regulation of negative emotions.

DETAILED DESCRIPTION:
Children and adolescents (herein "youths") treated in outpatient mental health care span a broad range of problems and disorders, with substantial comorbidity, and their most pressing problems and treatment needs may shift during treatment. These challenges may be addressed by treatment that is flexible and transdiagnostic (i.e., applicable to multiple mental health problems and disorders). A recent transdiagnostic treatment, FIRST, created in collaboration with community practitioners and intervention scientists, uses a principle-based approach to support efficient learning and implementation by clinicians. FIRST is built upon five empirically supported principles of change (e.g., calming, problem solving), each applicable to treatment of depression, anxiety/OCD, trauma, and misconduct. Three open benchmarking trials of FIRST, using low-cost clinician training and group consultation, have shown steep slopes of clinical improvement in youths treated in outpatient clinics.

This randomized controlled effectiveness trial will provide a more definitive test of FIRST, an initial investigation of a candidate mechanism of change, and tests of therapist characteristics that may predict and moderate implementation of evidence-based practices. The sample will be ethnically and economically diverse youths, ages 7-15, from four community clinics-two in greater Boston MA, two in greater Austin TX-all referred by their families and all showing elevated depression, anxiety/OCD, post-traumatic stress, or conduct problems. Clinicians within each clinic will be randomly assigned to learn and use FIRST or to employ Usual Care (UC), and youths will be randomized to FIRST or UC. Clinical outcomes will include change on standardized measures of mental health and on severity of the specific problems identified as most important by each youth and each caregiver at baseline. Study measures will include a proposed mechanism-regulation of negative emotions- thought to be responsive to treatment and responsible for changes in mental health. Analyses will assess whether treatment with FIRST impacts regulation, and whether improved regulation accounts for outcomes of FIRST treatment relative to UC. Finally, the study will investigate whether clinicians' baseline knowledge of, attitudes toward, and motivation to use evidence-based practices predicts or moderates their implementation of such practices in psychotherapy. The study will thus provide the first randomized trial of this new practice-adapted transdiagnostic treatment, plus an inquiry into the process through which it may work and therapist factors that may strengthen or weaken implementation.

ELIGIBILITY:
Inclusion Criteria:

* ages 7.0-15.9 years
* at least one clinically-relevant CBCL subscale score indicating borderline/clinical-range anxiety, depression, conduct problems, or post-traumatic stress
* English fluency indicated by taking all school classes in English

Exclusion Criteria:

* current suicide risk, operationalized as active suicidal ideation or a history of suicide attempt or inpatient hospitalization for suicide risk within the last 3 months
* presence of an eating disorder, schizophrenia spectrum disorder, autism spectrum disorder, or intellectual disability requiring special class placement in school
* referral for ADHD if specifically and exclusively to address inattentiveness and/or hyperactivity-impulsivity

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Child Behavior Checklist (CBCL; Achenbach & Rescorla, 2001) and Youth Self-Report (YSR; Achenbach & Rescorla, 2001) | Change from baseline to 18 months (quarterly at 0, 3, 6, 9, 12, and 18 months from 0 up to 78 weeks)
  The CBCL is a parent-report checklist with 113 youth problem items, each rated on a 0-1-2 scale (0 = not true, 1 = somewhat/sometimes true, 2 = very often true). The YSR is a corresponding 112-item youth-report checklist measure. From both the CBCL and the YSR, T-scores, adjusted for age and gender, Internalizing, Externalizing, and Total Problems scales will be used for outcome assessment. Higher scores represent more severe problems, with borderline and clinical cutoffs at T = 60 and T = 63, respectively. Evidence of CBCL/YSR validity and reliability is strong and extensive.
Behavior and Feelings Survey (BFS; Weisz et al., 2020) | Change from baseline through end of treatment (weekly from 0 up to 78 weeks)
  The 12-item BFS is a measure of internalizing (6 items), externalizing (6 items), and total problems, developed via four studies, three with samples of clinically referred youths aged 7-15 and their caregivers. Both youth and caregiver forms showed robust factor structure, internal consistency, test-retest reliability, convergent and discriminant validity in relation to three well-established symptom measures (including CBCL and YSR), and slopes of change indicating efficacy in monitoring treatment progress during therapy. Items are rated on a scale from 0 (not a problem) to 4 (a very big problem). Internalizing and externalizing scale scores range from 0 to 24 and total problems from 0 to 48 (with higher scores indicating greater problem severity).
Functional Top Problems Assessment (TPA; Weisz et al., 2011) | Change from baseline through end of treatment (weekly from 0 up to 78 weeks)
  The TPA assesses youth and caregiver severity ratings (from 0 = not a problem to 4 = a very big problem) for the functional top three problems the youth and caregiver independently identified as most important to them, in separate baseline interviews. Psychometric analyses have shown strong test-retest reliability, convergent and discriminant validity for the TPA in relation to standardized measures, and sensitivity to change during treatment.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule Short Form (PANAS-C/P-SF; Laurent et al., 1999; Ebesutani et al., 2011) | Change from baseline through end of treatment (weekly from 0 up to 78 weeks)
  Derived from the original Positive and Negative Affect Schedule, the brief 10-item PANAS includes 5 adjectives for positive affect (joyful, cheerful, happy, lively, proud) and 5 for negative affect (miserable, mad, afraid, scared, sad), on which youth and their parents report the extent to which they felt each on a 5- point Likert scale from 1 (very slightly or not at all) to 5 (extremely). Evidence of convergent and divergent validity of both the positive and negative affect scale scores with reports of anxiety and depressive symptoms has been found as well as good internal consistency of both scales. The 10-item version has shown similar validity and reliability properties and superior measurement properties as compared to the 27-item version. Total positive and negative affect scale scores range from 5 to 25, such that higher scores reflect stronger endorsement of positive or negative mood states.
Coping Questionnaire (CQ; Crane & Kendall, 2020) | Change from baseline through end of treatment (weekly from 0 up to 78 weeks)
  The CQ was developed in the context of the youth anxiety treatment research to assess youth and caregiver ratings of the youths' ability to regulate the emotional arousal associated with anxiety disorders. The CQ procedure is both idiographic (each youth and each caregiver identifies three situations that make the youth most upset) and standardized (each youth and each caregiver then rates, for each situation, the youth's ability "to make yourself (or himself/herself) feel less upset" on a 1 to 7 Likert scale). This simple measure, tested with a sample of 442 7-17 year-olds, showed good evidence of internal consistency, convergent and divergent validity in relation to measures of psychopathology and functioning, and criterion validity in its association with clinical severity ratings of the youths' principle diagnosis on a standardized diagnostic interview.
Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID parent version; Sheehan et al., 2010) | Change from baseline (0 months) to end of treatment (up to 78 weeks)
  The parent version of the MINI-KID is a structured diagnostic interview for DSM-IV and ICD-10 youth psychiatric disorders. It has been shown to provide efficient and highly reliable and valid diagnoses.
UCLA PTSD Reaction Index (PTSDRI; Steinberg et al., 2004) | Baseline for entire sample; quarterly (3, 6, 9, 12, and 18 months) for up to 18 months for those with elevated baseline PTS symptoms (from 0 up to 78 weeks)
  The PTSDRI has been widely used to assess PTS symptoms in children and teens. Various studies have shown good evidence of internal consistency, test-retest reliability, and validity relative to both degree of exposure to traumas and to PTSD diagnoses on standardized interviews.

OTHER OUTCOMES:
Evidence-Based Practice Attitudes Scale (EBPAS-15; Aarons, 2004) | Baseline
  Clinicians' EBP attitudes will be assessed using the EBPAS, which yields four subscales: appeal (EBP is intuitively appealing), requirements (would use EBP if required), openness (general openness to innovation), and divergence (perceived divergence between EBP and current practices). In a sample of 1,089 clinicians nested within 100 clinics in 75 cities in 26 states, internal consistency alpha was .76 for the total score, and ranged from .66 to .91 for the subscales. Confirmatory factor analyses support the theorized structure, with item loadings on the aforementioned scales ranging from 0.49 to 0.99, and these loading onto an overall attitudes towards EBP factor. The EBPAS openness scale is correlated with clinician report of CBT use, whereas the EBPAS divergence scale is correlated with clinician report of non-evidence-based strategies use.
Evidence-Based Treatment Intentions (EBTI; Williams, 2015) | Baseline
  The EBTI is designed to measure clinicians' intentions to adopt EBPs clinically. Derived from research on EBP adoption in youth service systems, the instructions define an EBP as ''a specific treatment protocol that has been developed through research and is supported by the results of controlled treatment studies.'' Sample item: ''Out of the next 10 new clients you see, how many would you expect to treat using an EBP?'' Internal consistency alpha for the scale was 0.80 in two studies with community clinicians.
Knowledge of Evidence Based Services Questionnaire (KEBS-Q; Stumpf et al., 2009) | Baseline, post-training (approx 2 weeks after training)
  The KEBSQ is a 40-item self-report measure of knowledge of practice elements in empirically supported and unsupported youth mental health treatments. Participants are asked to classify each item as included or not included in efficacious treatments for four problem areas (e.g., A = anxious/avoidant, D= depressed/withdrawn, B = disruptive behavior, H = hyperactivity, N = none). Scores have been shown to reliably distinguish between graduate students and practitioners, and to be sensitive to change after a half-day training in evidence-based practices. Each item is scored from 0 to 4, with one point assigned for each correct endorsement and one point for each correct rejection. Thus, total scores range from 0 to 160, with higher scores indicating more EBP knowledge.
Therapeutic Alliance Scale for Children and Caregivers/Parents(TASC-r; Shirk et al., 2011; TASCP; Accurso et al., 2013) | Monthly beginning after first session through end of treatment (every 4 weeks from 0 up to 78 weeks)
  The 12-item TASC-r and TASCP will be used to assess quality of the therapeutic alliance with the therapist, as reported by both youths and caregivers/parents, respectively. Items are rated a 4-point Likert scale (1 = not true; 4 = very true), with higher scores (ranging from 7 to 28) reflective of stronger alliance. Both have previously evidence good reliability and validity.
Therapy Process Observational Coding System-Alliance Scale (TPOCS-A; McLeod & Weisz, 2005) | Assessed throughout treatment via observational coding (ongoing from 0 up to 78 weeks)
  Youth-therapist and caregiver-therapist alliance will be assessed unobtrusively throughout treatment, using the TPOCS-A applied to recordings of therapy sessions. The TPOCS-A was derived from questionnaire measures of alliance, adapting items that could be observed directly, reflecting alliance (e.g., "demonstrates positive affect toward therapist," "work together equally on tasks") or its absence (e.g., "hostile toward therapist," "does not comply with tasks"). The measure was designed for clinical practice contexts. Psychometric analyses using youth and parent sessions in community outpatient clinics showed that both youth and parent forms have good inter-rater reliability (most intraclass correlation coefficients .50s - .60s), internal consistency (α = .95), associations with established youth- and parent-report questionnaire measures of alliance, and prediction of treatment outcome.
Therapist Satisfaction Index (TSI; Chorpita et al., 2015) | Immediately after treatment
  The TSI is a 16-item therapist-report measure on therapist attitudes toward manualized treatments. Psychometric analyses with youths treated in community clinics by 77 clinicians revealed two psychometrically sound subscales: perceived effectiveness (α = .82) and perceived responsiveness (α = .81). Items rated on a 5-point Likert scale (1 = strongly disagree; 5 = strongly agree), and higher total scores (ranging from 8 to 40 on each subscale) indicate greater satisfaction.
Parent and Child Satisfaction Scales (PCSS) | At first quarterly assessment after treatment ends (up to 78 weeks)
  The PCSS offers parallel parent- and youth-report measures of satisfaction with treatment. The parent measure (sample item: "Overall, how much progress did your child make in treatment at this clinic?") has shown good internal consistency (α = .85) and 7-14-day test-retest reliability (r = .83) in samples of parents of clinic-referred youths. The child measure (sample item: "Going to the clinic helped me with my problems") showed good internal consistency (α = .95) and 7-14-day test-retest reliability (r = .80) in samples of clinic-referred youths. Items are rated on a scale from 0 (very unhappy) to 4 (very happy), with greater total scores (ranging from 8 to 32) indicative of higher overall satisfaction.
Therapist Integrity in Evidence-Based Interventions (TIEBI; Jensen et al., 2004) | Assessed throughout treatment via observational coding (ongoing from 0 up to 78 weeks)
  Treatment sessions will be audio-recorded and coded for presence/absence of the evidence-based treatment procedures of FIRST, using a randomly selected 25% of FIRST and UC sessions. The TIEBI involves coding sessions in 5-minute segments for presence/absence of 27 items reflecting FIRST content, and coder ratings of therapist competence (skillfulness of delivery, rated from 0 to 4).
Engagement of families in treatment | Post-treatment (up to 78 weeks)
  Clinic records will provide detailed data on aspects of the treatment process related to engagement. These will include percent of scheduled sessions attended, attended on time, cancelled, and missed due to no-show; and, whether or not treatment was terminated as planned with therapist agreement.
Perceptions of Supervisory Support Scale (PSSS; Fukui et al., 2014) | Post-treatment (up to 78 weeks)
  The PSSS is a 22-item measure capturing the extent to which mental health providers feel supported in supervision. Items are rates on a 1 to 6 Likert scale (1 = never; 6 = always), with 6 indicating greater perceived supervisory support.
TCU Organizational Readiness for Change (TCU-ORC; Organizational Climate Scale; Institute of Behavioral Research, 2009) | Baseline
  The Organizational Climate Scale of the TCU ORC is a tool used to measure various components of an organization's institutional climate, including clarity of mission, cohesion, autonomy, communication, stress, and openness to change. The scale includes 30 items, which are rated on a 5-point Likert scale (1=strongly disagree; 5=strongly agree). Item scores are summed, such that higher scores represent stronger organizational climate.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Harvard University, Cambridge, Massachusetts
  - University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be uploaded to the NIMH Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be uploaded biannually per the NIH requirements starting in 2023. IPD will be available once the study findings are accepted for publication.
Access Criteria: - IPD can be accessed by scientific investigators by requesting data directly from the NDA. The NDA Data Access Committee will determine whether the proposed use of the dataset including the types of analyses is ethically appropriate and provide approval for researchers to access data uploaded to the NDA.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Cho E, Bearman SK, Woo R, Weisz JR, Hawley KM. A Second and Third Look at FIRST: Testing Adaptations of A Principle-Guided Youth Psychotherapy. J Clin Child Adolesc Psychol. 2021 Nov-Dec;50(6):919-932. doi: 10.1080/15374416.2020.1796678. Epub 2020 Aug 7. PMID 32762554
- [Background] Weisz J, Bearman SK, Santucci LC, Jensen-Doss A. Initial Test of a Principle-Guided Approach to Transdiagnostic Psychotherapy With Children and Adolescents. J Clin Child Adolesc Psychol. 2017 Jan-Feb;46(1):44-58. doi: 10.1080/15374416.2016.1163708. Epub 2016 Jul 21. PMID 27442352
- [Background] Weisz JR, Vaughn-Coaxum RA, Evans SC, Thomassin K, Hersh J, Ng MY, Lau N, Lee EH, Raftery-Helmer JN, Mair P. Efficient Monitoring of Treatment Response during Youth Psychotherapy: The Behavior and Feelings Survey. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):737-751. doi: 10.1080/15374416.2018.1547973. Epub 2019 Jan 18. PMID 30657721
- [Background] Weisz JR, Chorpita BF, Frye A, Ng MY, Lau N, Bearman SK, Ugueto AM, Langer DA, Hoagwood KE; Research Network on Youth Mental Health. Youth Top Problems: using idiographic, consumer-guided assessment to identify treatment needs and to track change during psychotherapy. J Consult Clin Psychol. 2011 Jun;79(3):369-80. doi: 10.1037/a0023307. PMID 21500888
- [Background] Laurent J, Catanzaro SJ, Joiner TE, Rudolph KD, Potter KI, Lambert S, Osborne L, Gathright T. A measure of positive and negative affect for children: Scale development and preliminary validation. Psychological Assessment. 1999; 11(3): 326-338.
- [Background] Ebesutani C, Okamura K, Higa-McMillan C, Chorpita BF. A psychometric analysis of the Positive and Negative Affect Schedule for Children-Parent Version in a school sample. Psychol Assess. 2011 Jun;23(2):406-16. doi: 10.1037/a0022057. PMID 21381834
- [Background] Daughters SB, Reynolds EK, MacPherson L, Kahler CW, Danielson CK, Zvolensky M, Lejuez CW. Distress tolerance and early adolescent externalizing and internalizing symptoms: the moderating role of gender and ethnicity. Behav Res Ther. 2009 Mar;47(3):198-205. doi: 10.1016/j.brat.2008.12.001. Epub 2008 Dec 13. PMID 19135649
- [Background] Crane ME, Kendall PC. Psychometric Evaluation of the Child and Parent Versions of the Coping Questionnaire. Child Psychiatry Hum Dev. 2020 Oct;51(5):709-720. doi: 10.1007/s10578-020-00975-w. PMID 32157488
- [Background] Aarons GA. Mental health provider attitudes toward adoption of evidence-based practice: the Evidence-Based Practice Attitude Scale (EBPAS). Ment Health Serv Res. 2004 Jun;6(2):61-74. doi: 10.1023/b:mhsr.0000024351.12294.65. PMID 15224451
- [Background] Steinberg AM, Brymer MJ, Decker KB, Pynoos RS. The University of California at Los Angeles Post-traumatic Stress Disorder Reaction Index. Curr Psychiatry Rep. 2004 Apr;6(2):96-100. doi: 10.1007/s11920-004-0048-2. PMID 15038911
- [Background] Williams NJ. Assessing mental health clinicians' intentions to adopt evidence-based treatments: reliability and validity testing of the evidence-based treatment intentions scale. Implement Sci. 2016 May 5;11:60. doi: 10.1186/s13012-016-0417-3. PMID 27150798
- [Background] Shirk SR, Karver MS, Brown R. The alliance in child and adolescent psychotherapy. Psychotherapy (Chic). 2011 Mar;48(1):17-24. doi: 10.1037/a0022181. PMID 21401270
- [Background] McLeod BD, Weisz JR. The therapy process observational coding system-alliance scale: measure characteristics and prediction of outcome in usual clinical practice. J Consult Clin Psychol. 2005 Apr;73(2):323-33. doi: 10.1037/0022-006X.73.2.323. PMID 15796640
- [Background] Lawson GM, Moore TM, Okamura KH, Becker-Haimes EM, Beidas RS. Knowledge of Evidence-Based Services Questionnaire: Development and Validation of a Short Form. Adm Policy Ment Health. 2020 Jul;47(4):581-596. doi: 10.1007/s10488-020-01020-7. PMID 32076887
- [Background] Chorpita BF, Park A, Tsai K, Korathu-Larson P, Higa-McMillan CK, Nakamura BJ, Weisz JR, Krull J; Research Network on Youth Mental Health. Balancing effectiveness with responsiveness: Therapist satisfaction across different treatment designs in the Child STEPs randomized effectiveness trial. J Consult Clin Psychol. 2015 Aug;83(4):709-18. doi: 10.1037/a0039301. Epub 2015 May 18. PMID 25984802
- [Background] Sheehan DV, Sheehan KH, Shytle RD, Janavs J, Bannon Y, Rogers JE, Milo KM, Stock SL, Wilkinson B. Reliability and validity of the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID). J Clin Psychiatry. 2010 Mar;71(3):313-26. doi: 10.4088/JCP.09m05305whi. PMID 20331933
- [Background] Fukui S, Rapp CA, Goscha R, Marty D, Ezell M. The perceptions of supervisory support scale. Adm Policy Ment Health. 2014 May;41(3):353-9. doi: 10.1007/s10488-013-0470-z. PMID 23377768
- [Background] Accurso EC, Hawley KM, Garland AF. Psychometric properties of the Therapeutic Alliance Scale for Caregivers and Parents. Psychol Assess. 2013 Mar;25(1):244-52. doi: 10.1037/a0030551. Epub 2012 Oct 22. PMID 23088205
- [Background] Institute of Behavioral Research. TCU Organizational Readiness for Change (ORC-D4). Fort Worth: Texas Christian University, Institute of Behavioral Research. 2009.
- [Derived] Bailin A, Cho E, Sternberg A, Evans SC, Hollinsaid NL, Bearman SK, Weisz JR. Principle-Guided Psychotherapy for Children and Adolescents (FIRST): study protocol for a randomized controlled effectiveness trial in outpatient clinics. Trials. 2023 Oct 21;24(1):682. doi: 10.1186/s13063-023-07717-y. PMID 37864269
- [Derived] Bailin A, Cho E, Sternberg A, Evans SC, Hollinsaid NL, Kate Bearman S, Weisz JR. Principle-Guided Psychotherapy for Children and Adolescents (FIRST): Study Protocol for a Randomized Controlled Effectiveness Trial in Outpatient Clinics. Res Sq [Preprint]. 2023 Sep 8:rs.3.rs-3210987. doi: 10.21203/rs.3.rs-3210987/v1. PMID 37720052